CLINICAL TRIAL: NCT03736343
Title: Individual Differences in the Effects of Alcohol (IDEA) Study
Brief Title: Impulsivity and Alcohol Response
Acronym: IDEA
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The COVID-19 outbreak began, precluding further participant recruitment for this protocol, which could only be conducted in-person. A decision was made that ample data was available to end data collection earlier than anticipated.
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); American Psychological Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB201801192 - N; OCR16172 (Other: Universiy of Florida); 5T32AA025877 (NIH)
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Use Disorder (AUD); Subjective Response to Alcohol (SR)
Keywords: impulsivity; family history; heavy drinking; blood alcohol content (BAC); breath alcohol content (BrAC)
MeSH Terms: conditions — Alcoholism; Impulsive Behavior | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Young Adult Heavy Drinkers Group 1 (Active Comparator): Young adult heavy drinkers, aged 21-30, will be administered varying doses of oral alcohol.
  Interventions: Drug: Alcohol
- Young Adult Heavy Drinkers Group 2 (Active Comparator): Young adult heavy drinkers, aged 21-30, will be administered varying doses of oral alcohol.
  Interventions: Drug: Alcohol

INTERVENTIONS:
Drug: Alcohol — Participants will complete two drinking sessions.
  Other Names: 80-proof Vodka Mixed Drinks

SUMMARY:
Impulsivity, a well-known risk factor predicting negative outcomes, refers broadly to a proclivity towards rapid action with a suboptimal regard for future consequences. Importantly, impulsivity is a multidimensional construct incorporating generalized and behavioral facets. However, underlying mechanisms linking facets of impulsivity to high-risk drinking remain uncertain. Such mechanisms, if uncovered, may be more appropriate intervention targets than impulsivity directly.

Similar to impulsivity, subjective response to alcohol (SR), or individual differences in sensitivity to the pharmacologic effects of alcohol, is an established risk factor for alcohol use disorder. Specifically, experiencing heightened rewarding stimulation and dampened aversive sedation from alcohol are related to high-risk drinking. Theory and recent findings indicate SR and impulsivity may be related, suggesting SR may be a mechanism linking facets of impulsivity to high-risk drinking. However, findings linking impulsivity to SR were all from secondary data analyses and most studies reported on only a single measure of impulsivity. For these reasons, an original data collection using laboratory alcohol administration methods is needed to address which facets of impulsivity are related to SR among young adult drinkers and whether these effects manifest while blood alcohol concentrations are increasing or declining.

This study will utilize a laboratory alcohol administration design to investigate whether distinct facets of impulsivity (i.e., generalized, choice, response) are related to subjective responses (i.e., stimulation and sedation) following alcohol administration.

DETAILED DESCRIPTION:
Young adult heavy drinkers, aged 21-30, will enroll in a laboratory alcohol administration study. In a simulated bar laboratory, participants will be administered oral alcohol with three vodka-based drinks. This procedure will allow collection of several measures, notably a widely used, validated measure of self-reported SR and multiple measures capturing facets of impulsive behavior prior to and following alcohol administration. Participants will be recruited through a number of means. Flyers will be posted and handed out in and around the various colleges, universities and technical schools in the Gainesville area as well as in other public areas. The study team will utilize the internet by posting brief solicitation messages on social media, newspaper sites, and classified advertising sites. These same brief messages will also be disseminated to students at the local colleges, universities and technical schools in the area via batch emails and list servs. When permitted, brief recruitment talks will be given verbally during class meetings at these local institutions. Verbal recruitment messages will contain the same material in the appended flyers and other advertisements. Copies of flyers will also be provided at the conclusion of these brief recruitment talks. Potential participants will complete an initial eligibility questionnaire over the phone or online. Participants who appear eligible based on the phone/web screen will be invited to attend an in-person screening appointment. If eligible, participants will be scheduled for two alcohol drinking sessions separated by a minimum of one and a maximum of seven days. After the second drinking session, participants will be scheduled for a follow-up appointment.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 21-30
* Be able to read English and complete study evaluations
* Drink alcohol regularly
* Be willing to consume vodka-based alcoholic beverages

Exclusion Criteria:

* Have positive urine screen results at the in-person screening or on the day of an alcohol drinking session for illegal drugs
* A woman who is pregnant, nursing, or refuses to use a reliable method of birth control.
* A current undergraduate or graduate student at any level in one of the departments that make up the College of Health and Human Performance (HHP) at the University of Florida (UF), where Dr. Leeman's faculty appointment is.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Biphasic Alcohol Effects Scale | Up to 6 hours
  Biphasic Alcohol Effects Scale is a 14-item, 2-factor model including stimulant and sedative alcohol effects. The minimum value for each of the 2 factors is 0 and the maximum is 70. Higher scores indicate greater stimulation and sedation for each factor, respectively.

SECONDARY OUTCOMES:
Subjective Effects of Alcohol Scale | Up to 6 hours
  The Subjective Effects of Alcohol Scale is a 14-item, 4-factor model including low and high arousal positive and negative alcohol effects. The current study assesses specifically high arousal negative (e.g., aggressive) and low arousal positive (e.g., relaxed) alcohol effects.The factor concerning high arousal negative alcohol effects ranges from 0 - 30, with higher scores indicating greater high arousal negative alcohol effects (e.g., aggression). The factor concerning low arousal positive alcohol effects ranges from 0 - 40, with higher scores indicating greater low arousal positive alcohol effects (e.g., relaxed).
Alcohol Reward | Up to 6 hours
  The Drug Effects Questionnaire will be used to assess the extent to which participants like the effects of alcohol they are experiencing at the time, rated on a 100-mm line (from "not at all" to "very much") and how much they want more alcohol at the time, also rated on a 100-mm line (from "not at all" to "very much").

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Principal Investigator — University of Florida
Locations (1):
- EDGE Lab, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No